CLINICAL TRIAL: NCT00495274
Title: A Single-centre, Open-label, Randomized, Single-dose, 6-way Crossover Study to Investigate the Pharmacokinetics, Safety and Tolerability of 6 Different Formulations of SB-649868 30 mg (Part A) and the Effect of Food on the Selected Formulation of SB-649868 Pharmacokinetic (Part B) in Healthy Male Volunteers
Brief Title: Bioequivalence and Food Effect Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OXS105205
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Bioequivalent; pharmacodynamic; Reference formulation; 5 new formulation; Food effect; Pharmacokinetics
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — N-((1-((5-(4-fluorophenyl)-2-methyl-4-thiazolyl)carbonyl)-2-piperidinyl)methyl)-4-benzofurancarboxamide; D-Worm; Granuflex E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy male subjects (Experimental): In Part A each subject will participate in six sessions and will be administered, in randomized order, single doses of five new formulations (formulation B, C, D, E and F) of SB-649868 30 milligrams (mg), in fasted state and a single dose of the original formulation (formulation A), after a standard Food and Drug Administration (FDA) High-Fat breakfast. All dosing sessions will be separated by a washout session of at least 5 ± 2 days after each dose. In Part B a single dose of the selected SB-649868 30 mg formulation will be administered after a standard FDA High-Fat breakfast.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Drug: Formulation F; Drug: Formulation G

INTERVENTIONS:
Drug: Formulation A — Formulation A represents the original formulation. SB-649868 10 mg film coated tablet (3 tablets to reach 30 mg), containing micronized drug substance. Formulation A will be administered in Part A.
  Other Names: SB-649868
Drug: Formulation B — Formulation B will represent SB-649868 10 mg film coated tablet containing micronized drug substance (3 tablets to reach 30 mg), but contains additional surfactant. Formulation B will be administered in Part A.
Drug: Formulation C — Formulation C will represent SB-649868 10 mg lipophilic capsule (3 capsules to reach 30 mg). Formulation C will be administered in Part A.
Drug: Formulation D — Formulation D will represent SB-649868 10 mg film coated tablet (3 tablets to reach 30 mg), containing nanomilled and spray dried powder. Formulation D will be administered in Part A.
Drug: Formulation E — Formulation E will represent SB-649868 10 mg capsule (3 capsules to reach 30 mg), containing nanomilled and spray dried powder. Formulation E will be administered in Part A.
Drug: Formulation F — Formulation F will represent SB-649868 15 mg liquid filled capsule (2 capsules to reach 30 mg). Formulation F will be administered in Part A.
Drug: Formulation G — Formulation G will be the selected formulation of SB-649868 30 mg to be assessed in Part B. The formulation will be administered after a standard FDA High-Fat breakfast

SUMMARY:
The purpose of this study is to select the formulation with the optimal pharmacokinetic profile for an hypnotic drug to further develop in the market.

DETAILED DESCRIPTION:
A single-centre, open-label, randomized, single-dose, 6-way crossover study to investigate the pharmacokinetics, safety and tolerability of 6 different formulations of SB-649868 30 mg (Part A) and the effect of food on the selected formulation of SB-649868 pharmacokinetic (Part B) in healthy male volunteers

ELIGIBILITY:
Inclusion criteria:

* Healthy adult male subjects aged between 18 and 65 years of age inclusive.
* Body weight and BMI within the protocol ranges.
* Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring.
* Circulating levels of LH, FSH and testosterone within the normal reference range.
* Signed and dated written informed consent.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion criteria:

* Positive pre-study urine drug screen and alcohol breath test.
* Positive pre-study Hepatitis B surface antigen, Hepatitis C antibody, or HIV ½ result.
* Abuse of alcohol as per protocol criteria.
* Consumption of prohibited food and drink as per protocol.
* Subject who is not prepared to eat the standard meals provided by the site.
* Use of prescription or non-prescription drugs 1 or 2 weeks before the first dose of study medication.
* Where participation in study would result in donation of blood in excess of 500mL within a 56 day period.
* History or presence of allergy to the study drug or drugs of this class, or a history of other allergy.
* Smoking history in the last three months as per protocol.
* An unwillingness of male subjects to follow contraception methods as per protocol.
* History or presence of significant psychiatric, respiratory or gastrointestinal illnesses, hepatic or renal diseases or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* The subject is unable or unwilling to abstain from strenuous physical activity in the 48 hours before screening and in the 48 hours before and the 48 hours after the treatment period.
* Current or previous (within 6 months) participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-07-02 (Actual); Primary Completion 2007-09-26 (Actual); Study Completion 2007-09-26 (Actual)

PRIMARY OUTCOMES:
-Part A: SB-649868 levels of 6 formulation predose, 0.5, 1, 1.5, 2,3,4,5,6,8,12 and 24hours post-dose | predose, 0.5, 1, 1.5, 2,3,4,5,6,8,12 and 24hours post-dose
-Part B: SB-649868 levels of selected formulation after food at the same timepoints as in Part A | predose, 0.5, 1, 1.5, 2,3,4,5,6,8,12 and 24hours post-dose

SECONDARY OUTCOMES:
-AE, Lab values and cardiovascular monitoring throughout study participation | throughout study participation
-Romberg heel-to-toe test at discharge | at discharge
-Cognitive functions predose, 0.5, 1, 2, 4, 6 hours post-dose | predose, 0.5, 1, 2, 4, 6 hours post-dose
Pharmacodynamic endpoint: Bond Lader Visual Analogue Scale (VAS) score | pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Verona, Veneto, Italy

REFERENCES:
- See also: Results for study OXS105205 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/OXS105205?search=study&search_terms=OXS105205#rs